CLINICAL TRIAL: NCT04648085
Title: Effect of Trigeminal Nerve Stimulation on Subbasal Corneal Nerve Plexus Density and Chronic Ocular Pain in Patients With Dry Eye
Brief Title: Effect of Trigeminal Nerve Stimulation on Corneal Nerves and Chronic Ocular Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CI-006-2020
Record Dates: First submitted 2020-11-21; First posted 2020-12-01 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Dry Eye; Neuropathic Pain; Eye Pain
Keywords: Transcutaneous Electric Stimulation; In vivo Confocal Microscopy; Subbasal Corneal Nerve Plexus; Dry Eye; Neuropathic Pain
MeSH Terms: conditions — Dry Eye Syndromes; Neuralgia; Eye Pain

STUDY DESIGN:
Intervention Model Description: Prospective, open, single-arm pilot study without randomization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Pre and Post Treatment with Trigeminal Nerve Stimulation (TNS) (Experimental): Individuals will receive treatment with trigeminal nerve stimulation for 20 minutes at a frequency of 100 Hertz (Hz). Ocular pain intensity will be recorded prior and after the use of therapy.
  Interventions: Device: Trigeminal Nerve Stimulation

INTERVENTIONS:
Device: Trigeminal Nerve Stimulation — Applied to to the forehead using a self-adhesive electrode positioned bilaterally over the upper branches of the trigeminal nerve.The device generates electrical impulses allowing to stimulate the trigeminal nerve.

SUMMARY:
Individuals with dry eye tend to present with ocular pain which persists despite the use of topical treatment. This could be secondary to somatosensory impairment attributable to neuropathic pain. The purpose of this study is to evaluate the effect of trigeminal nerve stimulation (TNS) on corneal nerves and chronic ocular pain in patients with dry eye.

DETAILED DESCRIPTION:
Dry eye is a multifactorial disease that produces a variety of clinical manifestations including, dryness, pain, blurred vision, and sensitivity to light or wind. Differences have been noted between the symptoms reported and the signs presented on physical examination, which suggests the involvement of somatosensory impairment. Ocular neuropathic pain is characterized by burning pain, hyperalgesia, photophobia, and sensitivity to wind. There are common physiopathological pathways, suggesting that corneal nerve sensitization contributes to the development of dry eye symptoms. Furthermore, in vivo confocal microscopy has reported a decrease in the density of the subbasal plexus in patients with a neuropathic component and dry eye, suggesting that they are not mutually exclusive conditions. Various topical treatments, as well as systemic medications are known to manage eye pain and dry eye. However, in some cases, individuals have been refractory to them, enhancing the importance of research in adjuvant therapies such as TNS.

This research protocol evaluates the effect of transcutaneous stimulation on corneal subbasal plexus density and chronic eye pain in patients with dry eye. A complete dry eye examination will be performed, including completion of Ocular Surface Disease Index (OSDI) and Dry Eye Questionnaire-5 (DEQ-5). Subbasal nerves density will be measured by confocal microscopy before and after receiving treatment with TNS. In addition, monthly monitoring of the intensity of ocular pain (with a numerical scale of 0-10) will be maintained. The intensity and severity of the clinical variables will be compared before and after receiving the treatment with a paired t-test considering a value of p<0.05 as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with dry eye, Ocular pain for more than 3 months, Contact lens users, Individuals using topical treatment and/or systemic medication for dry eye syndrome, Individuals with history of photo-ablative ocular surgery (Laser-assisted in situ keratomileusis (LASIK) , Photorefractive keratectomy (PRK), Small incision lenticule extraction(SMILE), Individuals with history of autoimmune disease (Lupus, Rheumatoid Arthritis, Sjögrens),

Exclusion Criteria:

* Individuals with pacemakers or implantable defibrillators, Individuals with diagnosis of epilepsy, History of facial trauma one month prior to recruitment, Acute facial pain with unknown etiology, History of ocular surgery one month prior to recruitment, Trigeminal neuralgia, Active Herpes Zoster Ophthalmicus,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Identify the effect of trigeminal nerve stimulation on chronic eye pain in patients with dry eye. | From three-six months
  Eye pain will be evaluated prior to the use of trigeminal nerve stimulation using a numeric pain scale ranging from 0-10, "0" indicating no pain and "10" indicating the most severe pain imaginable.
  Pain will be evaluated posterior to therapy with trigeminal nerve stimulation with the same scale during monthly follow up.
Identify the effect of trigeminal nerve stimulation on subbasal corneal nerve plexus density in patients with dry eye. | 2 months- 6 months
  Initial subbasal corneal nerve plexus density will be measured prior to therapy with with in vivo confocal microscopy.
  Density measurements will be repeated every two months with in vivo confocal microscopy posterior to trigeminal nerve stimulation use.

CONTACTS AND LOCATIONS:
Overall Officials: Simran Mangwani Mordani, MD, Principal Investigator — Instituto de Oftalmología Conde de Valenciana
Locations (1):
- Instituto de Oftalmología Conde de Valenciana, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Galor A, Moein HR, Lee C, Rodriguez A, Felix ER, Sarantopoulos KD, Levitt RC. Neuropathic pain and dry eye. Ocul Surf. 2018 Jan;16(1):31-44. doi: 10.1016/j.jtos.2017.10.001. Epub 2017 Oct 12. PMID 29031645
- [Background] Craig JP, Nelson JD, Azar DT, Belmonte C, Bron AJ, Chauhan SK, de Paiva CS, Gomes JAP, Hammitt KM, Jones L, Nichols JJ, Nichols KK, Novack GD, Stapleton FJ, Willcox MDP, Wolffsohn JS, Sullivan DA. TFOS DEWS II Report Executive Summary. Ocul Surf. 2017 Oct;15(4):802-812. doi: 10.1016/j.jtos.2017.08.003. Epub 2017 Aug 8. PMID 28797892
- [Background] De Paiva CS, Corrales RM, Villarreal AL, Farley WJ, Li DQ, Stern ME, Pflugfelder SC. Corticosteroid and doxycycline suppress MMP-9 and inflammatory cytokine expression, MAPK activation in the corneal epithelium in experimental dry eye. Exp Eye Res. 2006 Sep;83(3):526-35. doi: 10.1016/j.exer.2006.02.004. Epub 2006 Apr 27. PMID 16643899
- [Background] Karson CN, Burns RS, LeWitt PA, Foster NL, Newman RP. Blink rates and disorders of movement. Neurology. 1984 May;34(5):677-8. doi: 10.1212/wnl.34.5.677. PMID 6231489
- [Background] Dworkin RH, O'Connor AB, Kent J, Mackey SC, Raja SN, Stacey BR, Levy RM, Backonja M, Baron R, Harke H, Loeser JD, Treede RD, Turk DC, Wells CD. Interventional management of neuropathic pain: NeuPSIG recommendations. Pain. 2013 Nov;154(11):2249-2261. doi: 10.1016/j.pain.2013.06.004. Epub 2013 Jun 6. PMID 23748119
- [Background] Kalangara JP, Galor A, Levitt RC, Covington DB, McManus KT, Sarantopoulos CD, Felix ER. Characteristics of Ocular Pain Complaints in Patients With Idiopathic Dry Eye Symptoms. Eye Contact Lens. 2017 May;43(3):192-198. doi: 10.1097/ICL.0000000000000249. PMID 26925537
- [Background] Farhangi M, Feuer W, Galor A, Bouhassira D, Levitt RC, Sarantopoulos CD, Felix ER. Modification of the Neuropathic Pain Symptom Inventory for use in eye pain (NPSI-Eye). Pain. 2019 Jul;160(7):1541-1550. doi: 10.1097/j.pain.0000000000001552. PMID 30883524
- [Background] Woolf CJ, Salter MW. Neuronal plasticity: increasing the gain in pain. Science. 2000 Jun 9;288(5472):1765-9. doi: 10.1126/science.288.5472.1765. PMID 10846153
- [Background] Crane AM, Feuer W, Felix ER, Levitt RC, McClellan AL, Sarantopoulos KD, Galor A. Evidence of central sensitisation in those with dry eye symptoms and neuropathic-like ocular pain complaints: incomplete response to topical anaesthesia and generalised heightened sensitivity to evoked pain. Br J Ophthalmol. 2017 Sep;101(9):1238-1243. doi: 10.1136/bjophthalmol-2016-309658. Epub 2017 Jan 18. PMID 28100479
- [Background] Matsumoto Y, Ibrahim OMA. Application of In Vivo Confocal Microscopy in Dry Eye Disease. Invest Ophthalmol Vis Sci. 2018 Nov 1;59(14):DES41-DES47. doi: 10.1167/iovs.17-23602. PMID 30481805
- [Background] Tavakoli M, Hossain P, Malik RA. Clinical applications of corneal confocal microscopy. Clin Ophthalmol. 2008 Jun;2(2):435-45. doi: 10.2147/opth.s1490. PMID 19668734
- [Background] Zhang M, Chen J, Luo L, Xiao Q, Sun M, Liu Z. Altered corneal nerves in aqueous tear deficiency viewed by in vivo confocal microscopy. Cornea. 2005 Oct;24(7):818-24. doi: 10.1097/01.ico.0000154402.01710.95. PMID 16160498
- [Background] Alhatem A, Cavalcanti B, Hamrah P. In vivo confocal microscopy in dry eye disease and related conditions. Semin Ophthalmol. 2012 Sep-Nov;27(5-6):138-48. doi: 10.3109/08820538.2012.711416. PMID 23163268
- [Background] Kinard KI, Smith AG, Singleton JR, Lessard MK, Katz BJ, Warner JE, Crum AV, Mifflin MD, Brennan KC, Digre KB. Chronic migraine is associated with reduced corneal nerve fiber density and symptoms of dry eye. Headache. 2015 Apr;55(4):543-9. doi: 10.1111/head.12547. Epub 2015 Mar 31. PMID 25828778
- [Background] Aggarwal S, Kheirkhah A, Cavalcanti BM, Cruzat A, Colon C, Brown E, Borsook D, Pruss H, Hamrah P. Autologous Serum Tears for Treatment of Photoallodynia in Patients with Corneal Neuropathy: Efficacy and Evaluation with In Vivo Confocal Microscopy. Ocul Surf. 2015 Jul;13(3):250-62. doi: 10.1016/j.jtos.2015.01.005. Epub 2015 Feb 20. PMID 26045233
- [Background] Small LR, Galor A, Felix ER, Horn DB, Levitt RC, Sarantopoulos CD. Oral Gabapentinoids and Nerve Blocks for the Treatment of Chronic Ocular Pain. Eye Contact Lens. 2020 May;46(3):174-181. doi: 10.1097/ICL.0000000000000630. PMID 31206369
- [Background] Sivanesan E, Levitt RC, Sarantopoulos CD, Patin D, Galor A. Noninvasive Electrical Stimulation for the Treatment of Chronic Ocular Pain and Photophobia. Neuromodulation. 2018 Dec;21(8):727-734. doi: 10.1111/ner.12742. Epub 2017 Dec 28. PMID 29283468
- [Background] Noseda R, Burstein R. Migraine pathophysiology: anatomy of the trigeminovascular pathway and associated neurological symptoms, cortical spreading depression, sensitization, and modulation of pain. Pain. 2013 Dec;154 Suppl 1:S44-53. doi: 10.1016/j.pain.2013.07.021. Epub 2013 Jul 25. PMID 23891892
- [Background] Zayan K, Aggarwal S, Felix E, Levitt R, Sarantopoulos K, Galor A. Transcutaneous Electrical Nerve Stimulation for the Long-Term Treatment of Ocular Pain. Neuromodulation. 2020 Aug;23(6):871-877. doi: 10.1111/ner.13146. Epub 2020 Mar 20. PMID 32196838
- [Background] Martinez JD, Galor A, Ramos-Betancourt N, Lisker-Cervantes A, Beltran F, Ozorno-Zarate J, Sanchez-Huerta V, Torres-Vera MA, Hernandez-Quintela E. Frequency and risk factors associated with dry eye in patients attending a tertiary care ophthalmology center in Mexico City. Clin Ophthalmol. 2016 Jul 21;10:1335-42. doi: 10.2147/OPTH.S106451. eCollection 2016. PMID 27499613
- [Background] Galor A, Feuer W, Lee DJ, Florez H, Venincasa VD, Perez VL. Ocular surface parameters in older male veterans. Invest Ophthalmol Vis Sci. 2013 Feb 19;54(2):1426-33. doi: 10.1167/iovs.12-10819. PMID 23385801
- [Background] Patel DV, McGhee CN. Mapping of the normal human corneal sub-Basal nerve plexus by in vivo laser scanning confocal microscopy. Invest Ophthalmol Vis Sci. 2005 Dec;46(12):4485-8. doi: 10.1167/iovs.05-0794. PMID 16303938